CLINICAL TRIAL: NCT03351673
Title: Endometrial Volume as a Predictor of Endometrial Pathology in Perimenopausal Uterine Bleeding Endometrial Volume as a Predictor of Endometrial Pathology in Perimenopausal Uterine Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hanan Nabil, Assistant Professor, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Endometrial volume
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Endometrial Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endometrial volume 2D TVS (Experimental): perimenopausal women who bleed are examined by 2D TVS and the calculated endometrial volume using a specific formula and followed by endometrial biopsy for correlation with the pathological findings
  Interventions: Diagnostic Test: endometrial volume 2D TVS

INTERVENTIONS:
Diagnostic Test: endometrial volume 2D TVS — calculation the endometrial volume using 2D ultrasound and correlation the results with the pathological findings of endometrial biopsy

SUMMARY:
Endometrial thickness has been used as an indicator of risk for endometrial hyperplasia and carcinoma in asymptomatic perimenopausal women. However, there is no cutoff value in perimenopausal women and the same thickness does not express the same endometrial volume in different endometrium because uterine lengths may be different and endometrial irregularities may exist. Many studies assessed endometrial volume measured by three-dimensional (3D) TVS as a predictor of malignancy in women with postmenopausal bleeding. To our knowledge there is no study assess endometrial volume measured by two dimension TVS in prediction of endometrial pathology, however it is cheap and available than 3D TVS.

ELIGIBILITY:
Inclusion Criteria:

*perimenopausal women with abnormal bleeding e.g. menorrhagia, metrorrhagia and polymenorrhea.

Exclusion Criteria:

*general or local causes of bleeding, drug intake or recent hormonal contraception

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
accuracy of measurement of endometrial volume by 2D TVS in prediction of endometrial pathology | 1year

CONTACTS AND LOCATIONS:
Locations (1):
- mansoura University, Al Mansurah, Dakahlia Governorate, Egypt